CLINICAL TRIAL: NCT00144183
Title: An Open-label Study Evaluating the Resistance Profile of Single Dose Nevirapine(NVP) When Combined With a 4 or 7 Day Course of Combivir® (ZDV/3TC) Compared to Single Dose Nevirapine for the Prevention of Mother to Child Transmission (pMTCT) of HIV - Treatment Options Preservation Study (T.O.P.S.)
Brief Title: A Study of Single Dose Nevirapine (NVP) Combined With Combivir® for the Prevention of Mother to Child Transmission (pMTCT) - Treatment Options Preservation Study (TOPS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1100.1413; MCC;N2/19/8/2(1958)
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Nevirapine; Zidovudine

INTERVENTIONS:
Drug: Nevirapine (NVP) — Nevirapine 200mg once daily for 14 days followed by 200mg twice daily thereafter for the remainder of the treatment period. Combivir®, one tablet twice daily.
Drug: Zidovudine (ZCV)
Drug: 3TC

SUMMARY:
To determine whether a regimen of single dose nevirapine combined with either 4 or 7 days of Combivir®, compared to a regimen of single dose nevirapine, for the prevention of mother to child transmission can reduce the rate of development of drug resistant mutations of HIV-1, in HIV-1 infected pregnant women, who have not received antiretroviral therapy previously.

DETAILED DESCRIPTION:
An open-label, randomised, multicentre study to determine whether a regimen of single dose nevirapine combined with either 4 or 7 days of Combivir, compared to a regimen of single dose nevirapine, for the prevention of mother to child transmission can reduce the rate of development of drug resistant mutations of HIV-1, in HIV-1 infected pregnant women, who have not received antiretroviral therapy previously.

An interim analysis of the first 61 patients showed that a clinical and statistical difference exists between the occurrence of HIV-1 NNRTI resistant mutations in the single dose nevirapine only arm (50%) and the two other combination arms (9%). These findings partially answered the objectives outlined in the initial objectives. Consequently enrolment onto the single dose nevirapine arm was terminated. The objective of the trial was modified to compare whether either the 4 or the 7 day combination of ZDV+3TC and nevirapine would result in any significant reduction in the incidence of nevirapine resistance.

Study Hypothesis:

Evaluations of HIV-1 resistance patterns in trials of pMTCT have demonstrated nevirapine resistant HIV-1 isolates in approximately 15-20% of mothers 4-6 weeks after receiving either a single or two dose 200mg nevirapine regimen. Although the ability to detect these genotypic mutations decreases to 0% by about 18 months, it is not clear whether this resistance is clinically significant.(HIVNET 012).

Empirically then it would seem useful to develop a strategy to diminish the emergence of this early resistance, therefore this study is proposed to evaluate whether the effect of 4 or 7 days of 3TC+ ZDV added to a single dose nevirapine regimen for the prevention of MTCT will prevent the emergence of resistance to nevirapine.

Comparison(s):

ACTG 076, Thai, PETRA , HIVNET 006/012, SAINT

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women identified at antenatal clinics after from 34 weeks gestation and who are antiretroviral drug naive.
* Mothers with a documented positive HIV Rapid test confirmed by a detectable HI V-1 RNA PCR (viral load).
* Mother to have a screening viral load of > 2000 RNA copies/mL.

Exclusion Criteria:

* Mothers who, in the opinion of the investigator ,cannot be relied on to return with their infants for postnatal visits.
* Mothers who have received any antiretroviral drugs previously.
* Clinical suspicion of intra-uterine foetal death
* Unwillingness or inability to reasonably comply with the protocol requirements.
* Use of any other investigational product during the pregnancy and for the dura tion of the study period.
* Patients with a recent history of pancreatitis or peripheral neuropathy.
* Patients with renal failure requiring dialysis.
* Patients with evidence of hepatic dysfunction as measured by total bilirubin > 2.5 times ULN or AST/ALT > 5 times ULN at the screening visit.
* Patients with any one of the following additional laboratory abnormalities at screening : Haemoglobin concentration < 7.5 g/dl. Neutrophil count < 750 cells/mm3. Platelet count < 75,000 cells/mm3. Serum amylase > 2 x ULN.
* recent history ( during the pregnancy) of drug abuse or alcoholism.
* Mothers who will undergo elective caesarean section.
* If known prior to delivery, mothers with foetuses with anomalies incompatible with life.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407
Dates: Start 2003-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01

PRIMARY OUTCOMES:
Percentage of mothers with HIV-1 isolates with new NNRTI (Non Nucleoside Reverse Transcriptase Inhibitor) resistance-associated mutations identified by genotype testing | 6 weeks following delivery

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. South Africa (Pty.) Ltd.
Locations (5):
- South Africa (5):
  - Boehringer Ingelheim Investigational Site, Attridgeville
  - Boehringer Ingelheim Investigational Site, Cape Town
  - Boehringer Ingelheim Investigational Site, Durban
  - Boehringer Ingelheim Investigational Site, Johannesburg
  - Boehringer Ingelheim Investigational Site, Soweto

REFERENCES:
- [Derived] McIntyre JA, Hopley M, Moodley D, Eklund M, Gray GE, Hall DB, Robinson P, Mayers D, Martinson NA. Efficacy of short-course AZT plus 3TC to reduce nevirapine resistance in the prevention of mother-to-child HIV transmission: a randomized clinical trial. PLoS Med. 2009 Oct;6(10):e1000172. doi: 10.1371/journal.pmed.1000172. Epub 2009 Oct 27. PMID 19859531